CLINICAL TRIAL: NCT04395898
Title: Pancreaticoduodenectomy: Outcomes of a Complex Surgical Procedure From a Developing Country
Status: Completed | Type: Observational
Sponsor: Shaukat Khanum Memorial Cancer Hospital & Research Centre (Other)
Responsible Party: Principal Investigator, aun jamal, Fellow in Surgical Oncology, Shaukat Khanum Memorial Cancer Hospital & Research Centre
Other Study IDs: EX-24-10-19-01
Record Dates: First submitted 2020-05-11; First posted 2020-05-20 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Pancreaticoduodenectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: pancreaticoduodenectomy — Whipple's procedure

SUMMARY:
ABSTRACT

BACKGROUND Pancreaticoduodenectomy (PD) plays an integral part in the management of pancreatic, periampullary and duodenal cancers along with few other pathologies of this region. Despite advances in surgery PD continues to have significant morbidity and noteworthy mortality. The aim of this study is to provide an in-depth report on the patient characteristics, indications and the outcomes of PD) in a tertiary cancer hospital in Pakistan.

MATERIALS AND METHODS:

The study population included patients who underwent PD between January 1st 2014 and march 31st 2019, at Shaukat Khanum Memorial Cancer Hospital and Research Centre (SKMCH&RC) in Pakistan. The Data was retrospectively analyzed from the Hospital Information System (HIS), which is a prospectively maintained patient electronic database of SKMCH&RC. Patient characteristics, procedural details and post-operative outcomes according to internationally accepted definitions were reported.

KEYWORDS: Whipple's procedure, Pancreaticoduodenectomy, Pancreaticogastrostomy, lower middle income, pancreatic fistula, periampullary cancer.

DETAILED DESCRIPTION:
INTRODUCTION:

Pancreatic cancer is one of the most common cancer worldwide and ranks 7th as the leading cause of death among all cancers.The estimated 5 year survival of pancreatic cancer is very poor i.e. 5%. Apart from cancer there is a plethora of benign and pre-malignant pancreatic lesions that can manifest symptoms in patients.

Surgery plays an integral part in the management of pancreatic lesions. Pancreaticoduodenectomy (PD) is a considered to be one of the most complex and morbid surgical procedures. The first case series published by Allan Whipple in 1935 reported the procedure related mortality in excess of 25 percent. With the advancements in surgical techniques, perioperative and critical care management, mortality rate has dropped down to less than 5 percent in high volume centers. However, morbidity remains high with some studies reporting up to 70 percent .

There have been some studies, with small cohort and limited follow up periods, reporting on outcomes of PD in Pakistan .To our knowledge, no published study has focused on detailed surgical outcomes and long term follow up. We do not know the long term outcomes after PD in Pakistan and most information is based on a western literature which may not be applicable to a Pakistani cohort of patients. SKMCH&RC being a dedicated cancer centre and tertiary care hospital of the country receives a high number of referrals of patients requiring this complex procedure in Pakistan.

Every patient that is referred to our hospital has a detailed history and examination in the walk-in clinic. Every case undergoes a pancreatic protocol Computerised Tomograph scan(CT) and where appropriate interventions like Endoscopic Retrograde Cholangiography (ERCP) with or without stent placement, Endoscopic Ultra-sound or Percutaneous Trans-hepatic Cholangiogram (PTC) are undertaken. Every case is discussed in our Multi-Disciplinary Team (MDT) meeting comprising of trained hepatobiliary surgeons, gastroenterologists, diagnostic and interventional radiologists, pathologists, medical and radiation oncologists. Patients with border-line operable confirmed pancreatic cancers undergo neo-adjuvant treatment, whereas resectable lesions undergo upfront PD.investigators work at a paperless hospital and all patient data is put real time into a computerised Hospital Information System (HIS) by all cadres including nurses, allied health professionals and doctors. The hospital has a unique in-house developed computerised patient management system (HIS) that collects all patient information in real time including patient demographics, investigations, Multi-Disciplinary Team discussions, Nursing assessments, outpatient, operative notes and post- operative outcomes. As the data is collected in real time and stored, it allows for accurate retrospective review of the data.

The aim of this study is to provide a detailed analysis of the patient characteristics, indications, post-operative and intermediate term outcomes for PD in a Pakistani cohort of patients. This will provide a reference point for physicians when they counsel their patients regarding PD outcomes in Pakistan and also help define areas of potential improvement in the future.

METHODOLOGY:

Patients:

All patients undergoing PD from 1st January 2014 till 31st March 2019 at SKMCH&RC, Pakistan were retrospectively evaluated from a prospectively maintained database using the HIS system. The cohort of patients selected included malignant, pre-malignant and benign pathologies. Exclusion criteria included patients that did not undergo PD after exploratory laparotomy due to metastatic disease or with involvement of celiac, superior mesenteric or hepatic arteries. The ethical approval was sought from Institutional Review Board (IRB) of SKMCH & RC vide number EX-24-10-19-01.

Variables:

Variables recorded were age, gender, co-morbidities, American-Society of Anesthesiologists score (ASA), pre-operative histopathology, clinical staging, surgical details, post-operative complications, mortality (30 & 90 day), length of stay, and survival outcomes.

Pancreatic fistula was recorded as defined by ISGPF 2016 updated criteria. Post-Pancreatectomy Hemorrhage (PPH) was recorded as defined by International Study Group on Pancreatic Surgery (ISGPS) 2007 classification. Morbidity was recorded according to Clavien-Dindo classification.

Statistical analyses:

Calculations were performed with Statistical Package for the Social Sciences (SPSS Ver20) for Windows. Data was described using median with minimum and maximum value for skewly distributed quantitative variables. For categorical variables, number of observations and percentages were reported. For survival analyses Kaplan-Miere Curve was applied. The study is in compliance with the SKMCH&RC guidelines on research involving human subjects.

ETHICAL APPROVAL:

Ethical approval was obtained from Institutional Review Board (IRB) of Shaukat Khanum Memorial Cancer Hospital and Research Centre, prior to the commencement of study.

PATIENTS' CONSENT:

Informed consent was taken from every patient about data collection, analysis and research publication.

DECLARATIONS OF INTEREST:

None

FUNDING:

The research did not receive any specific grant from funding agencies in the public, commercial, or not-for-profit sectors.

ELIGIBILITY:
Inclusion Criteria:

all patients whose surgeries were done from January 2014 to March 2019

Exclusion Criteria:

None as such

Ages: 19 Years to 78 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Pancreatic cancer.
Sampling Method: Non-Probability Sample
Enrollment: 161 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Survival analysis | 4 years
  disease free and overall survival

SECONDARY OUTCOMES:
Morbidity | 30 days
  morbidity was defined according to Clavien-Dindo classification
recurrence | 4 years
  recurrence is defined as return of the cancer after initial curative or definitive treatment, can be local or distant

CONTACTS AND LOCATIONS:
Overall Officials: Farah Rasheed, Study Director — Clinical research officer
Locations (1):
- Shaukat Khanam Memorial Cancer Hospital and Research Center, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
will see
Supporting Information: Study Protocol
Time Frame: will see
Access Criteria: that will be discussed with the hospital IRB and later we will see wether it has to be shared